CLINICAL TRIAL: NCT03295071
Title: Observational Registry Study of Leber Hereditary Optic Neuropathy (LHON) Affected Patients
Brief Title: REALITY LHON Registry
Acronym: REALITY
Status: Completed | Type: Observational
Sponsor: GenSight Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: GS010_Registry_001
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-07

CONDITIONS: Leber Hereditary Optic Neuropathy
Keywords: Heredity Optic Atrophy; Leber Hereditary Optic Atrophy; Leber Hereditary Optic Neuropathy; Eye Diseases; Hereditary Eye Diseases; Inherited retinal dystrophies or degeneration; Inborn Genetic Disease; Gene Therapy; Intravitreal Injections; Mitochondrial Disease; AAV2 Vectors; Nervous System Diseases; Neurodegenerative Disease; Heredodegenerative Disorders of the Nervous System
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber; Eye Diseases; Eye Diseases, Hereditary; Genetic Diseases, Inborn; Mitochondrial Diseases; Nervous System Diseases; Neurodegenerative Diseases | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-group study: This study is a multi-country retrospective and cross-sectional observational study of affected LHON subjects, based on retrospective subjects' medical chart abstractions and cross-sectional administration of patient-reported outcomes (PROs).
  Interventions: Other: Patient-reported outcomes (PROs)

INTERVENTIONS:
Other: Patient-reported outcomes (PROs) — Patient-reported outcomes (PROs)

SUMMARY:
This study is a multi-country retrospective and cross-sectional observational study of affected LHON subjects, based on retrospective subjects' medical chart abstractions and cross-sectional administration of patient-reported outcomes (PROs).

DETAILED DESCRIPTION:
The purpose of this study is to understand the evolution of visual functional and structural changes and other associated symptoms in patients with LHON. The relation between genetic, lifestyle and/or environmental factors and the LHON disease will be described, and a better understanding of the natural history of LHON disease and the healthcare associated to with the disease will be sought.

In addition, we would also like to understand the economic burden for patients and their families with LHON resulting from direct and indirect costs they may have because of their disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a confirmed and genotyped diagnosis of LHON;
* Subjects with visual function outcomes data including at least 2 visual function assessments between 1 year and 3 years (+/- 4 weeks) after vision loss;
* Subjects who are willing and able to provide written informed consent if required as per local regulations;
* For LHON subjects under the age of 18 years, permission from a legal guardian to participate in the study;

Exclusion Criteria:

* Subjects who received any investigational drug, or participated in any LHON-related interventional clinical trial during the observational period;
* Subjects without medical charts data available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit at least 50 affected LHON subjects (both adult and pediatric) from global clinical sites at the following countries, but not limited to: Spain, Italy, France, United Kingdom, and the United States. Efforts will be done to maintain the population of at least 50 affected LHON subjects.
  Recruitment efforts of recruiting approximately 75% of eligible subjects with 11778/ND4 mutation and 30% of eligible subjects under the age of 18 at the time of index date, wherever possible, will be done at the study level.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Visual Function | All assessments available before enrollment
  Visual function will include visual examination data from medical records.
The National Eye Institute Visual Function Questionnaire (VFQ)-25 | Enrollment
  The National Eye Institute Visual Function Questionnaire (NEI-VFQ or VFQ)-25 is a valid and reliable 25-item version of the 51-item VFQ.
The 36-Item Short Form Health Survey (SF-36) | Enrollment
  The SF-36 surveys health status and quality of life
Child Health Questionnaire (CHQ) | Enrollment
  The CHQ uses the same structure and methodological approach as the SF-36 and is designed and normed for children from 5-to-18 years of age.
EuroQol-5 Dimension (EQ-5D)-5L | Enrollment
  The EuroQol-5 Dimension-5 Level (EQ-5D-5L) is a generic HRQoL instrument that is widely used as a PRO measure.

SECONDARY OUTCOMES:
Economic burden of disease | Enrollment
  Data will be gathered by questionnaire at cross-sectional survey. Direct costs and indirect costs resulting from LHON will be estimated by all enrolled subjects. Direct costs will include the medical and non-medical direct costs due to LHON

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - Doheny Eye Center UCLA Pasadena, Pasadena, California
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Wills Eye Institute, Philadelphia, Pennsylvania
  - Alkek Eye Center, Houston, Texas
- France (2):
  - CHU d'Angers, Angers
  - CHNO Les Quinze Vingts, Paris
- Italy (2):
  - Ospedale Bellaria, Bologna
  - Ospedale San Raffaele, Milan
- Institut Catala de Retina, Barcelona, Spain
- Moorfields Eye Hospital, London, Greater London, United Kingdom

REFERENCES:
- [Derived] Carelli V, Newman NJ, Yu-Wai-Man P, Biousse V, Moster ML, Subramanian PS, Vignal-Clermont C, Wang AG, Donahue SP, Leroy BP, Sergott RC, Klopstock T, Sadun AA, Rebolleda Fernandez G, Chwalisz BK, Banik R, Girmens JF, La Morgia C, DeBusk AA, Jurkute N, Priglinger C, Karanjia R, Josse C, Salzmann J, Montestruc F, Roux M, Taiel M, Sahel JA; the LHON Study Group. Indirect Comparison of Lenadogene Nolparvovec Gene Therapy Versus Natural History in Patients with Leber Hereditary Optic Neuropathy Carrying the m.11778G>A MT-ND4 Mutation. Ophthalmol Ther. 2023 Feb;12(1):401-429. doi: 10.1007/s40123-022-00611-x. Epub 2022 Nov 30. PMID 36449262
- [Derived] Newman NJ, Yu-Wai-Man P, Carelli V, Biousse V, Moster ML, Vignal-Clermont C, Sergott RC, Klopstock T, Sadun AA, Girmens JF, La Morgia C, DeBusk AA, Jurkute N, Priglinger C, Karanjia R, Josse C, Salzmann J, Montestruc F, Roux M, Taiel M, Sahel JA. Intravitreal Gene Therapy vs. Natural History in Patients With Leber Hereditary Optic Neuropathy Carrying the m.11778G>A ND4 Mutation: Systematic Review and Indirect Comparison. Front Neurol. 2021 May 24;12:662838. doi: 10.3389/fneur.2021.662838. eCollection 2021. PMID 34108929
- See also: GenSight Biologics Website — http://www.gensight-biologics.com/